CLINICAL TRIAL: NCT03038178
Title: An Open-label Study of Efficacy, Safety and Tolerability of Liposomal Amikacin for Inhalation (LAI) Once Daily in Addition to Standard Multi-antibiotic Therapy in the Treatment of Mycobacterium Abscessus Lung Disease
Brief Title: Liposomal Amikacin for Inhalation (LAI) in the Treatment of Mycobacterium Abscessus Lung Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kevin Winthrop (Other)
Collaborators: Insmed Incorporated (Industry); The University of Texas Health Science Center at Tyler (Other)
Responsible Party: Sponsor-Investigator, Kevin Winthrop, Associate Professor, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAI/INS-IIR-01
Record Dates: First submitted 2017-01-03; First posted 2017-01-31 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Mycobacterium Infections, Nontuberculous; Mycobacteria, Atypical
Keywords: Mycobacterium Infections, Nontuberculous; Mycobacteria, Atypical; Amikacin; Inhalation
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous; Mycobacterium Infections; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LAI plus multi-drug regimen (Experimental): once daily dosing of Liposomal-Amikacin for Inhalation (LAI) 590 mg for 12 months plus standard of care (SOC) mycobacterial multi-drug regimen in accordance with the 2007 ATS/ IDSA guidelines
  Interventions: Drug: LAI plus multi-drug regimen

INTERVENTIONS:
Drug: LAI plus multi-drug regimen — Liposomal Amikacin for Inhalation (LAI) is the experimental treatment which, in this single arm will be taken in conjunction with standard of care multi-drug treatment regimen
  Other Names: ARIKAYCE™

SUMMARY:
The proposed study will assess the efficacy, safety and tolerability of once daily dosing of Liposomal-Amikacin for Inhalation (LAI) 590 mg for 12 months plus standard of care (SOC) mycobacterial multi-drug regimen in accordance with the 2007 ATS/ IDSA guidelines, for treatment of mycobacterium abscessus lung disease.

DETAILED DESCRIPTION:
This is an open-label study of efficacy, safety and tolerability of once daily dosing of Liposomal-Amikacin for Inhalation (LAI), in addition to a standard multi-drug antibiotic therapy in accordance with the 2007 ATS/ IDSA guidelines, in patients with Mycobacterium abscessus lung disease. The multi-drug therapy is determined at the discretion of the Investigator. After screening, all eligible patients will enter the trial and will receive LAI 590 mg once daily for 12 months. If deemed necessary by the investigator, dose may be adjusted from a minimum of three times per week up to daily, in cases of adverse events relating to tolerability.

All patients who enter the study will have subsequent study visits at Months 1,2,4,6,9, at End-of-Study or Month 12, and at 1 and 3 months post study drug discontinuation. At each visit (including screening), review of concomitant medications, review of adverse events, and physical exam, will be performed. Chest CT scan will be performed at baseline, 6 months, and 12 months, unless a chest CT scan has already been performed within 6 months on this time point. The 6 minute walk test and QOL-B-NTM will be performed at baseline, 6 months, 12 months, and 3 months post study drug discontinuation. All patients will have inducted sputum collected at each study visit, and patients will self-collect expectorated sputum during intervening monthly time-points until study completion to determine changes in mycobacterial smear and culture status.

Unscheduled visits will occur as needed should subjects' symptoms worsen between visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 12 years and older
* Diagnosis of M. abscessus, including all subspecies, abscessus, bolleti, and massiliense lung disease according to the 2007 ATS/IDSA criteria
* Both newly diagnosed and currently on treatment or previously treated patients will be included
* Culture positive (either sputum or bronchoscopy) for M. abscessus at time of screening
* Willingness to adhere to a treatment regimen, study visits, and study procedures during the course of the study.
* Ability to produce at approximately 3.0 mL of sputum or be willing to undergo an induction that produces approximately 3.0 mL of sputum for culture collection
* Female of childbearing potential agrees to practice an acceptable method of birth control (e.g., abstinence, hormonal or barrier methods, partner sterilization, or IUD)
* Written informed consent or assent obtained from the patient, parent or legal guardian prior to the performance of any study related procedures

Exclusion Criteria:

* Active pulmonary tuberculosis requiring treatment at screening
* Treatment with inhaled or intravenous Amikacin within 14 days prior to baseline
* Known hypersensitivity to aminoglycosides
* Aspartate aminotransferase or alanine aminotransferase ≥ 3 times the upper limit of normal or total bilirubin ≥ 2 times the upper limit of normal (ULN) at screening
* Current addiction to alcohol or illicit drug abuse
* Any condition which in the opinion of the Investigator interferes with ability to adhere to study requirements
* Primary immunodeficiency syndromes and acquired immunodeficiency syndromes (e.g., HIV-positive patients regardless of CD4 counts)
* Absolute neutrophil count ≤500/μL at Screening
* Significant (as determined by the investigator) hearing loss, vestibular dysfunction, neuromuscular weakness or a diagnosis of myasthenia gravis, where the potential risk of aminoglycoside toxicity outweighs the potential benefit
* Serum creatinine >2 times ULN at Screening
* History of lung transplantation
* Any condition that, in the judgment of the Investigator, would compromise the ability of the subject to complete the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline sputum culture at 12 months | Sputum examined for culture change from Baseline at 12 months

SECONDARY OUTCOMES:
Change from Baseline 6-minute Walk Test at 6 months | 6-minute Walk Test results examined for change from Baseline at 6 months
Change from Baseline 6-minute Walk Test at 12 months | 6-minute Walk Test results examined for change from Baseline at 12 months
Change from End of Treatment (EOT) sputum culture at 3 months post EOT | Sputum examined for culture change from EOT at 3 months post EOT
Number of Hospitalizations for pulmonary exacerbations | Number of Hospitalizations for pulmonary exacerbations that occur between Baseline and 12 months
Number of Adverse Events | Number of Patient-reported and Investigator-reported Adverse Events at 12 months
Number of subjects discontinuing study drug due to Adverse Event | Number of subjects who discontinue study drug before 12 months due to Adverse Event will be examined at 12 months

OTHER OUTCOMES:
Change from Baseline reported nontuberculous mycobacterium (NTM) symptoms at End of Treatment (EOT) | Patient-reported NTM symptoms examined for change from Baseline at EOT (12 months)
Change from Baseline Chest CT at End of Treatment (EOT) | CT scan examined for change from Baseline at EOT (12 months)
Change from Baseline body weight at End of Treatment (EOT) | body weight of patient examined for change from Baseline at EOT (12 months)
Change from Baseline Body Mass Index (BMI) at End of Treatment (EOT) | BMI of patient examined for change from Baseline at EOT (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Winthrop, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - University of Texas Health Science Center, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siegel SAR, Griffith DE, Philley JV, Brown-Elliott BA, Brunton AE, Sullivan PE, Fuss C, Strnad L, Wallace RJ Jr, Winthrop KL. Open-Label Trial of Amikacin Liposome Inhalation Suspension in Mycobacterium abscessus Lung Disease. Chest. 2023 Oct;164(4):846-859. doi: 10.1016/j.chest.2023.05.036. Epub 2023 Jun 17. PMID 37419144